CLINICAL TRIAL: NCT00939562
Title: An Open-Label, Two-Treatment, Two-Period, Randomized Cross-Over Study To Assess The Bioequivalence Between Commercial Doxycycline Carragenate And Monohydrate Tablet Formulations In Normal Healthy Male Subjects
Brief Title: Bioequivalence Between Two Tablet Formulations Of Doxycycline Carragenate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A1901003
Record Dates: First submitted 2009-07-08; First posted 2009-07-15 (Estimated); Results first posted 2009-12-23 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-11

CONDITIONS: Bacterial Infection
Keywords: Bioequivalence
MeSH Terms: conditions — Bacterial Infections | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- doxycycline monohydrate tablet (Experimental)
  Interventions: Drug: doxycycline monohydrate tablet
- doxycycline carragenate tablet (Active Comparator)
  Interventions: Drug: doxycycline carragenate tablet

INTERVENTIONS:
Drug: doxycycline monohydrate tablet — Tablet, 100 mg, Single dose
  Arms: doxycycline monohydrate tablet
Drug: doxycycline carragenate tablet — Tablet, 100 mg, Single dose
  Arms: doxycycline carragenate tablet

SUMMARY:
The purpose of this protocol is to study if two different tablet formulations of doxycycline are bioequivalent to each other.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years.
* Body Mass Index (BMI) of 18 to 30 kg/m2.

Exclusion Criteria:

* Evidence or history of clinically significant abnormality.
* Any condition possibly affecting drug absorption.
* A positive urine drug screen.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Ahmedabad, Gujarat, India

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1901003&StudyName=Bioequivalence%20Between%20Two%20Tablet%20Formulations%20Of%20Doxycycline%20Carragenate

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxycycline Monohydrate, Then Doxycycline Carragenate: Single dose of one 100 mg doxycycline monohydrate tablet (Test) during first period and single dose of one 100 mg doxycycline carragenate tablet (Reference) during the second period.
- Doxycycline Carragenate, Then Doxycycline Monohydrate: Single dose of one 100 mg doxycycline carragenate tablet (Reference) during first period and single dose of one 100 mg doxycycline monohydrate tablet (Test) during the second period.
Period: Period 1
Arm/Group | Doxycycline Monohydrate, Then Doxycycline Carragenate | Doxycycline Carragenate, Then Doxycycline Monohydrate
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Doxycycline Monohydrate, Then Doxycycline Carragenate | Doxycycline Carragenate, Then Doxycycline Monohydrate
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes subjects who received a single dose of one 100 mg doxycycline monohydrate tablet (Test) and a single dose of one 100 mg doxycycline carragenate tablet (Reference).
Arm/Group | Entire Study Population
Number analyzed (Participants) | 24
Age, Customized [Number; unit: participants]
  < 18 years | 0
  18 to 44 years | 24
  45 to 64 years | 0
  > = 65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Doxycycline
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours postdose.
Population: The pharmacokinetic (PK) concentration population was defined as all subjects randomized and treated who had at least 1 concentration in at least 1 treatment period.
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- Doxycycline Monohydrate: Single dose of one 100 mg doxycycline monohydrate tablet (Test).
- Doxycycline Carragenate: Single dose of one 100 mg doxycycline carragenate tablet (Reference).
Arm/Group | Doxycycline Monohydrate | Doxycycline Carragenate
Number analyzed (Participants) | 24 | 24
ug/mL | 2.526 (0.5090) | 2.442 (0.4585)
Statistical Analysis 1: Comparison: Doxycycline Monohydrate vs Doxycycline Carragenate; Natural log transformed Cmax was analyzed using a mixed effects model (sequence, period and treatment were fixed effects and subject within sequence was a random effect); Test type: Superiority or Other; Ratio = 102.95, 90% CI [94.74 to 111.86] — The adjusted mean differences and 90% confidence intervals (CIs) were exponentiated to provide the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Doxycycline carragenate=Reference, doxycycline monohydrate=Test

2. Primary Outcome: Area Under Plasma Concentration-Time Profile From Time Zero to Infinity (AUCinf) of Doxycycline
Description: AUCinf = Area under the plasma concentration-time profile from time zero (pre-dose) to infinity.
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours postdose.
Population: PK
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Arm/Group | Doxycycline Monohydrate | Doxycycline Carragenate
Number analyzed (Participants) | 24 | 24
ug*hr/mL | 56.297 (10.3348) | 54.026 (11.4855)
Statistical Analysis 1: Comparison: Doxycycline Monohydrate vs Doxycycline Carragenate; Natural log transformed AUCinf was analyzed using a mixed effects model (sequence, period and treatment were fixed effects and subject within sequence was a random effect); Test type: Superiority or Other; Ratio = 104.67, 90% CI [98.95 to 110.73] — The adjusted mean differences and 90% CIs were exponentiated to provide the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Doxycycline carragenate=Reference, doxycycline monohydrate=Test

ADVERSE EVENTS:
Arm/Group | Doxycycline Monohydrate | Doxycycline Carragenate
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 1/24 | 2/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxycycline Monohydrate (N=24) | Doxycycline Carragenate (N=24)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.